CLINICAL TRIAL: NCT03823976
Title: A Pattern of Dental Treatment and Oral Rehabilitation for Adult Individuals With Intellectual Disability in General Anaesthesia
Brief Title: Dental Treatment and Oral Rehabilitation for Adult Individuals With Intellectual Disability in General Anaesthesia
Acronym: DTADGA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Novi Sad (Other)
Responsible Party: Principal Investigator, Bojan Petrovic, Principal Investigator, University of Novi Sad
Other Study IDs: 01454/2018
Record Dates: First submitted 2019-01-20; First posted 2019-01-31 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Intellectual Disabilities (F70-F79)
Keywords: dental care; oral rehabilitation; general anaesthesia; tooth loss
MeSH Terms: conditions — Intellectual Disability; Tooth Loss | interventions — Anesthesia, General

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Types of the dental procedures in general anaesthesia — Analysis of the mean number of preventive, prophylactic, therapeutic and rehabilitation procedures

SUMMARY:
This study evaluates the types of dental procedures performed in general anaesthesia for adult persons with intellectual disability, as well as factors affecting the decision to perform the dental treatment in general anaesthesia, factors contributing to tooth loss and possibilities to perform oral rehabilitation procedures

DETAILED DESCRIPTION:
Oral diseases are not life threatening and dental procedures usually do not pose significant risk to a patient. In situation where a patient does not tolerate dental treatment, and consequently general anaethesia (GA) is used, an intellectually disabled (ID) patient with a condition that is routinely managed in the general population is exposed to significantly higher medical risk. Quality of oral health care delivery for adults with ID is considered inadequate and in need of constant improvement. Therefore, the present study aims to analyse the type of dental treatment performed in GA and factors affecting the treatment. By its design this is an observational, epidemiological, retrospective study. A representative sample of the target population is realised by the assessment of approximately n=250 ID adults treated at the Dental Clinic of Vojvodina. A number of parameters such as severity of ID, the presence of concomitant conditions, living arrangements, medical diagnoses, physical status according to the American Society of Anesthesiologists' classification (ASA score), history of previous surgical/GA treatments and injuries/trauma, frequency of dental visits, procedures that were conducted in GA and during routine dental treatment (RDT), dental status including DMFT (decay, missed, filled teeth index) and total number of extracted teeth and data about oral rehabilitation.The use of GA emphasizes the inequalities in persons with ID, since it is always more radical compared to RDT. It is a frequent occurrence that with the use of GA only prevention of complications and pain relief are accomplished, resulting in a multiple teeth extractions. This approach inevitably leads to further dysfunctions in cranio-facial system, affecting all aspects of everyday life in persons with ID.

ELIGIBILITY:
Inclusion Criteria:

* Participants with ID older than 18 years at the time of treatment in GA
* Participants who had at least one general anesthesia dental treatment.

Exclusion Criteria:

* Participants who had dental treatment in GA due to physical condition, without ID
* Participants younger than 18,
* Participants with ID who had never had treatment in GA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study includes all patients older than 18 years that have been treated in general anesthesia between 2008 and 2018 at the Dentistry Clinic of Vojvodina, Serbia. Study gathered data from medical documentation of procedures which was obtained patient's/parents'/caregivers' consent for.
Sampling Method: Non-Probability Sample
Enrollment: 274 (Estimated)
Dates: Start 2019-01-20 (Actual); Primary Completion 2019-04-20 (Estimated); Study Completion 2019-06-20 (Estimated)

PRIMARY OUTCOMES:
Tooth loss analysis calculated as T fraction in DMFT teeth after the procedure | 3 months
  The analysis of the mean number of extracted teeth per patient during dental procedure in general anaesthesia. Correlations (odds-ratios) between the level of ID, the presence of comorbidities, institutionalisation and tooth loss
Oral rehabilitation analysis calculated as care index (CI), defined as the number of restored teeth as a fraction of the total number of decayed (D), missing (M) and filled (F) teeth (CI= F/DMF × 100). | 6months
  The analysis of oral rehabilitation procedures performed during general anaesthesia.Correlations (odds-ratios) between the level of ID, the presence of comorbidities, institutionalisation and the level of CI

CONTACTS AND LOCATIONS:
Overall Officials: Bojan B Petrovic, PhD, Principal Investigator — Faculty of Medicine, Dental Clinic of Vojvodina
Locations (1):
- Dental Clinic of Vojvodina, Novi Sad, Serbia

IPD SHARING:
Plan to Share IPD: Undecided